CLINICAL TRIAL: NCT02415764
Title: OnTrack>An Online Role-Playing Game: A Small Business Innovation Research (SBIR) Grant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R43MH105013-01 (NIH)
Record Dates: First submitted 2015-03-30; First posted 2015-04-14 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Psychosis; Schizoaffective Disorder; Schizophrenia
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pilot test Intervention OnTrack>The Game (Other): Consumers who have been referred to OnTrackNY sites at Washington Heights Community Service or Mental Health Association Westchester in the past six months will be recruited to participate in a product evaluation of OnTrack>The Game.
  Intervention: This is a behavioral/attitudinal intervention, using OnTrack>The Game, which will include each participant sitting down at a computer for approximately one hour (over the course of one week) to complete the prototype game. Users will take on the role of a person who has experienced first-episode psychosis and moves through animated role-playing scenarios, learn practical tips for engaging in care, play mini-games to develop self-advocacy skills, and view stories of hope and recovery (brief video vignettes).
  Interventions: Behavioral: Behavioral/Attitudinal OnTrack Role-Playing Game

INTERVENTIONS:
Behavioral: Behavioral/Attitudinal OnTrack Role-Playing Game — The intervention will involve each participant sitting down at a computer for approximately one hour (over the course of one week) to complete the prototype game. Users will take on the role of a person who has experienced first-episode psychosis and moves through animated role-playing scenarios, learn practical tips for engaging in care, play mini-games to develop self-advocacy skills, and view stories of hope and recovery (brief video vignettes).
  While the intervention does not require direct supervision by the research team, technical support will be available for the duration of the study via telephone, instant messaging and email. All participants receive identical baseline surveys and 2-week follow up surveys.

SUMMARY:
Our team will develop a prototype game (OnTrack>The Game) in which users play the role of a person who has experienced First Episode Psychosis and move through animated role-playing scenarios, learning practical tips for engaging in care, playing mini-games to develop self- advocacy skills, and seeing stories of hope and recovery (brief video vignettes). The game is designed in an engaging comic book style in which the player is presented with realistic situations designed to promote engagement and the development of trusting relationships.

Following development of the prototype, the investigators will conduct a pilot study to develop preliminary data to determine feasibility of a large-scale Phase 2 effectiveness study. This pilot study aims to demonstrate proof of concept for OnTrack>The Game. The investigators will recruit a sample of patients/consumers (n=25) from OnTrackNY sites that offer services for those experiencing their first psychotic episode. Quantitative data will be collected through baseline and follow up surveys that utilize instruments to measure knowledge and attitudes about recovery, perceptions of stigma, feelings of empowerment and sense of hopefulness. The investigators will also conduct semi-structured interviews with a subset of participants to explore engagement in treatment and attitudes toward the game.

DETAILED DESCRIPTION:
In light of research supporting early first episode psychosis (FEP) intervention models as well as the efficacy of video gaming to engage young people with FEP in treatment, the connection between the two needs to be explored. A gaming tool for first-episode psychosis has the potential to improve patient care; and, decrease stigma associated with schizophrenia.

Hypothesis:

The investigators hypothesize that Phase 1 of this study will demonstrate that the videogame is comprehensible, engaging and easy to maneuver. The investigators hypothesize that the results from the pilot study will suggest that this technologically innovative tool has potential to enhance positive outcomes of research-tested interventions, such as OnTrackNY, for individuals with FEP.

Approach:

Our team will develop a prototype game (OnTrack>The Game) in which users play the role of a person who has experienced FEP and move through animated role-playing scenarios, learning practical tips for engaging in care, playing mini-games to develop self- advocacy skills, and seeing stories of hope and recovery (brief video vignettes). The game is designed in an engaging comic book style in which the player is presented with realistic situations designed to promote engagement and the development of trusting relationships.

Following development of the prototype, the investigators will conduct a pilot study to develop preliminary data to determine feasibility of a large-scale Phase 2 effectiveness study. This pilot study aims to demonstrate proof of concept for OnTrack>The Game. The investigators will recruit a sample of patients/consumers (n=25) from OnTrackNY sites that offer services for those experiencing their first psychotic episode. Quantitative data will be collected through baseline and follow up surveys that utilize instruments to measure knowledge and attitudes about recovery, perceptions of stigma, feelings of empowerment and sense of hopefulness. The investigators will also conduct semi-structured interviews with a subset of participants to explore engagement in treatment and attitudes toward the game.

ELIGIBILITY:
Inclusion Criteria (Consumers):

* 18 - 30 years of age;
* have experienced a first episode of psychosis;
* have been referred to OnTrack New York in the past 12 months;
* are willing to complete study requirements; and
* provides informed consent

Exclusion Criteria (Consumers):

* non-English speaker;
* not clinically stable (at risk of self harming or others, and/or experiencing elevated symptoms) and incapable of providing informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Changes in attitudes toward recovery | Pre and post game play; timeframe: Months 9 and 10 (weeks 36 and 40)
  The Herth Hope Index (HHI) will be employed to assess hope in adults immediately before (Month 9; week 36) and 2 weeks (Month 10; week 40) following game play. The instrument is a 12-item survey adapted from the Herth Hope Scale (HHS) (Herth, 1992). The Recovery Attitudes Questionnaire (RAQ-16) will also be used, which helps consumers identify and think about their beliefs and attitudes toward recovery. The instrument is a 16-item survey that will be employed immediately before (week 36) and 2 weeks after game play (week 40) (Borkin et al, 2000).

SECONDARY OUTCOMES:
Sense of stigma and empowerment | Month 10 (week 40)
  (1) The self-stigma of mental illness survey (short form) (Corrigan et al, 2012) and (2) empowerment survey will be used both immediately before game play (weeks 36) and 2-weeks (week 40) following game play (Rogers, 1997).
Increased engagement in treatment | Post game play; timeframe: Month 10 (week 40)
  Semi-structured interviews will be conducted with a subset of participants to explore access to treatment and potential barriers.
Attitudes toward the game | Post game play; timeframe: Month 10 (week 40)
  Semi-structured interviews will take place with a subset of participants to explore their experience playing the game and attitudes toward it (e.g. extent to which they can relate to it; satisfaction; usability).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olivet, MA, Principal Investigator — Center for Social Innovation
Locations (2):
- United States (2):
  - Center for Social Innovation, Needham, Massachusetts
  - New York State Psychiatric Institute, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borkin, J. R., Stefffen, J. J., Ensfield, K. K., Wishnick, H., Wilder, K. & Yangarber, N. (2000) Recovery attitudes questionnaire: Development and evaluation. Psychiatric Rehabilitation Journal, 24(2), 95-102
- [Background] Corrigan PW, Michaels PJ, Vega E, Gause M, Watson AC, Rusch N. Self-stigma of mental illness scale--short form: reliability and validity. Psychiatry Res. 2012 Aug 30;199(1):65-9. doi: 10.1016/j.psychres.2012.04.009. Epub 2012 May 10. PMID 22578819
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Rogers ES, Chamberlin J, Ellison ML, Crean T. A consumer-constructed scale to measure empowerment among users of mental health services. Psychiatr Serv. 1997 Aug;48(8):1042-7. doi: 10.1176/ps.48.8.1042. PMID 9255837